CLINICAL TRIAL: NCT00878267
Title: A Qualitative Study of Patient-Reported Outcomes (PRO)-Based Palliative and Hospice Care Practice: Integrating PROs and Decision Support Into an Electronic Record
Brief Title: Patient-Reported Outcomes (PRO)-Based Palliative and Hospice Care Practice: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0840
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Cancer
Keywords: Cancer; Computer Program; Palliative Care; Patient-Reported Outcomes; PRO; Palliative and Hospice Care Practice; Electronic Health Record; EHR; Interview
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interview
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — 3 step process including person to person meeting and questionnaires taking about 30 minutes.
  Other Names: Survey

SUMMARY:
The goal of this research study is to collect information to plan how to design a computer program for cancer patients receiving palliative care, their caregivers, and doctors and nurses who work in palliative care. Researchers want to learn how to make this program practical for use by future patients, caregivers, doctors, and nurses.

DETAILED DESCRIPTION:
The Computer Program:

In this study, researchers will interview cancer patients receiving palliative care, their caregivers, and doctors and nurses who work in palliative care.

The computer program will be designed to help doctors and nurses monitor the symptoms of patients. The program will also be designed to help doctors and nurses make decisions about how to care for patients.

Interview Session:

If you agree to take part in this study, you will be interviewed by a research staff member. The study chair may also attend the interview. The interview will be held at the Palliative Care outpatient clinic.

The interview session will be done in 3 steps, which are described below. Each step will take about 10 minutes.

First, you will read questionnaires about patient symptoms. These questionnaires are drafts of the ones that will be included in the software program.

You will then look at a draft of the computer program's layout.

Last, you will be interviewed. You will be asked to discuss your experiences as a patient or caregiver in reporting symptoms and health status to doctors and nurses. You will also be asked to discuss what might make the program more usable.

During the interview, you may also be asked to answer sample questions on the draft questionnaires and discuss how readable you think the questions are. For example, you will discuss your opinion about the font size, text placement, and color scheme.

Study Data:

The interview session will be audio-taped. To protect your confidentiality, only your first name will be used during the interview session. Patients and their caregivers will also be interviewed separately to protect privacy.

Patient responses will not be disclosed to caregivers, and caregiver responses will not be disclosed to patients. The patient's palliative care doctor will be told, however, if patients or caregivers show signs of emotional difficulties.

When the audio recording is transcribed (typed) by the research staff, all names will be coded so that no one can be identified by name. The audio recordings will be stored in password-protected files that are available only to the study chair and staff.

After the results of the study are published, the audio recordings will be destroyed by the study staff.

Length of Study:

Your study participation will be over after the interview session.

This is an investigational study.

Up to 26 participants will be enrolled in this study. This includes up to 9 patients and 9 caregivers in this part of the study, and up to 4 doctors and 4 nurses in a second part of the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patient/caregiver participants will be adults 21 years of age or older.
2. Patient participants will be palliative care cancer patients and their caregivers.
3. Participating patients should be receiving palliative care at the MD Anderson Cancer Center.
4. Patient must be able to speak, read and write English
5. Physician and nurse experts in palliative care will be eligible for participation on the study's expert panel. (For study purposes, a physician or nurse expert is defined as a physician or nurse with a minimum of four years experience working in a palliative care setting.
6. Physician and nurse experts will be eligible for participation in study interviews if they have a minimum of four years experience working in a palliative care setting.

Exclusion Criteria:

1. Patients who are not able to self-report their symptom status using either paper-and-pencil or electronic tools.
2. Patients or caregivers who do not agree to sign the study's informed consent document.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UT MD Anderson Cancer Center (MDACC) cancer patients, 21 years of age or older, receiving palliative care, their caregivers, and UT MDACC physicians and nurses who work in palliative care.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Define Patient-Reported Outcomes (PRO)-based Palliative/Hospice Care Model Integrating PRO Results with Evidence-based Treatment Guidelines and Pathways to Care | 2 Years
  Through focused interviews with specific tasks: review PRO domains and questionnaires for the care mode; review user interface design and work flow; discuss user expectations of the system to assess the usability of a system's user interface design.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Kallen, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org